CLINICAL TRIAL: NCT04212234
Title: Echography in Pregnant Obese Women and Ultrasound Speed.
Brief Title: Pregnant Obese Women and Fetal Ultrasound Quality.
Acronym: EPOWUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: PHRC IR 2018 DELABAERE; 2018-A03478-47 (Other: ANSM)
Record Dates: First submitted 2019-08-30; First posted 2019-12-26 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Obese Women; Pregnant Women
Keywords: fetal ultrasound; ultrasound propagation velocity; image quality; obese women

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Scans will be evaluated by independent experts who had not performed the exams. Scans will be anonymized and ultrasound propagation velocity will not be reported on the images.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- free ultrasound propagation velocity (Experimental): ultrasound exams will be performed using several ultrasound propagation velocities
  Interventions: Device: ultrasound propagation velocities, ultrasound fetal quality
- conventional ultrasound propagation velocity (No Intervention): ultrasound exams will be performed using the 1540m/s conventional celerity

INTERVENTIONS:
Device: ultrasound propagation velocities, ultrasound fetal quality — Obese pregnant women will be included before the second trimester fetal ultrasound examination.
  Women will be allocated to one intervention group or to the control group. In the intervention group, the ultrasonographer will be able to use several ultrasound propagation velocities to perform the exam.
  In the control group, exam will be performed using the conventional ultrasound velocity.
  An exam will be considered to be complete if all the images recommended by national guideline are acquired. If ultrasound images are missing, other ultrasound exams may be performed until completeness is reached.
  The protocol will be applied for the second and the third fetal ultrasound examination which are recommended by national guideline.
  All scans will be evaluated by two independent experts who do not have performed any of the exams. They will evaluate the completeness of each exam. Each scan will be quoted using the quality score proposed by Salomon et al.
  Arms: free ultrasound propagation velocity

SUMMARY:
Ultrasound (US) image construction uses equations that contain the value of the propagation velocity of sound waves; this velocity is assumed conventionally to be constant and equal to 1540 m/s in the human body. Since 1977, all manufacturers of US scanners have used this value, which was first established in 1950. In fatty tissue, however, the actual propagation velocity is only in the order of 1450 m/s. US velocity in fat tissue is slower than in other soft tissues (ie:1450 m/s vs 1540 m/s) therefore the intrinsic image quality in terms of sharpness and precision is improved when considering this parameter for image construction The main objective of this study is to evaluate the impact of ultrasound propagation velocity setting on completeness of ultrasound exams and images quality during the second and third trimester fetal ultrasound examination in obese patients.

DETAILED DESCRIPTION:
Obese pregnant women will be included before the second trimester fetal ultrasound examination.

Women will be allocated to one intervention group or to the control group. In the intervention group, the ultrasonographer will be able to use several ultrasound propagation velocities to perform the exam.

In the control group, exam will be performed using the conventional ultrasound velocity.

An exam will be considered to be complete if all the images recommended by national guideline are acquired. If ultrasound images are missing, other ultrasound exams may be performed until completeness is reached.

The protocol will be applied for the second and the third fetal ultrasound examination which are recommended by national guideline.

All scans will be evaluated by two independent experts who do not have performed any of the exams. They will evaluate the completeness of each exam. Each scan will be quoted using the quality score proposed by Salomon et al.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index>30
* Between 20 and 25 weeks of gestation

Exclusion Criteria:

* Multiple pregnancy
* Uterine scare

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 596 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2024-10-19 (Actual); Study Completion 2024-10-19 (Actual)

PRIMARY OUTCOMES:
image quality of fetal ultrasound exam | second trimester and third trimester ultrasound exam
  Quality will be assessed by calculating Salomon's score for each image.
completeness of fetal ultrasound exam | second trimester and third trimester ultrasound exam
  completeness will be assessed by the number of the recommended images which could have been registered during the first ultrasound exam in each trimester.

SECONDARY OUTCOMES:
use of supplementary ultrasound exams in order to assess completeness | through study completion, an average of 1 year
  description of each modality of supplemental ultrasound exam
description of ultrasonographist method in order to improve ultrasound exam | through study completion, an average of 1 year
  description of modality
economic analysis of the intervention | through study completion, an average of 1 year
  cost-effectiveness analysis

CONTACTS AND LOCATIONS:
Overall Officials: Amélie Delabaere, MD, PhD, Principal Investigator — CHU de Clermont-Ferrand
Locations (5):
- France (5):
  - Hôpital Estaing - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Hôpital de la Croix Rousse - Hospices Civils de Lyon, Lyon
  - Hôpital Femme Mére Enfant - Hospices Civils de Lyon, Lyon
  - Hôpital Arnaud de Villeneuve - CHU de Montpellier, Montpellier
  - Hôpital Cochin - Assistance Publique - Hôpitaux de Paris, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Delabaere A, Chauveau B, Lemery D, Ollier A, Guiguet-Auclair C, Mourgues C, Legrand A. Protocol for the e-POWUS Project: multicentre blinded-randomised controlled trial of ultrasound speed choice to improve sonography quality in pregnant women with obesity. BMJ Open. 2021 Sep 21;11(9):e038684. doi: 10.1136/bmjopen-2020-038684. PMID 34548341